CLINICAL TRIAL: NCT02668484
Title: Randomized Comparison of Repositionable and Balloon-Expandable Prostheses in Patients Undergoing Trans-catheter Aortic Valve Implantation
Brief Title: REpositionable Versus BallOOn-expandable Prosthesis for Trans-catheter Aortic Valve Implantation
Acronym: REBOOT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LMU Klinikum (Other)
Responsible Party: Principal Investigator, Prof. Dr. Julinda Mehilli, Director, Interventional Cardiology, LMU Klinikum
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GEMucS001-15
Record Dates: First submitted 2016-01-26; First posted 2016-01-29 (Estimated); Last update posted 2019-06-03 (Actual); Status verified 2019-05

CONDITIONS: Aortic Valve Disease
Keywords: TAVI; trans-femoral; Sapien; Lotus
MeSH Terms: conditions — Aortic Valve Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- repositionable valve prosthesis (Experimental): Lotus
  Interventions: Device: repositionable valve prosthesis
- balloon-expandable valve prosthesis (Active Comparator): Sapien
  Interventions: Device: balloon-expandable valve prosthesis

INTERVENTIONS:
Device: repositionable valve prosthesis — repositionable valve prosthesis implanted via trans-femoral and trans-catheter route
  Other Names: Lotus
  Arms: repositionable valve prosthesis
Device: balloon-expandable valve prosthesis — balloon-expandable valve prosthesis implanted via trans-femoral and trans-catheter route
  Other Names: Sapien
  Arms: balloon-expandable valve prosthesis

SUMMARY:
There are different aortic valve prosthesis used for treatment of aortic valve disease through catheter-based procedures. The current study aims to compare two different aortic valve prosthesis regarding their outcomes at 30-day and 2-year follow-up.

DETAILED DESCRIPTION:
Important improvements in aortic valve prostheses technology has been made aiming comparable performance of these prosthesis to surgical valve ones.

The experience with the early generation of aortic valve prostheses revealed some important differences regarding the incidence of paravalvular leakage, need for pacemaker or valve thrombosis among them. Currently the new generations of valve prostheses such as Sapien 3 balloon-expandable valve and Lotus, repositionable valve are the most frequently used devices. There are registry data about the clinical performance of these valve types but a randomized comparison is missing.

ELIGIBILITY:
Inclusion Criteria:

1. Symptomatic aortic valve disease in need of valve replacement
2. Heart team (including at least a cardiac surgeon and an interventional cardiologist) agrees on the eligibility that trans-femoral TAVI is appropriate.
3. Study patient is an adult of legal consent age.
4. Study patient has provided written informed consent to participate in the study

Exclusion Criteria:

1. Life expectancy < 12 months due to co-morbid conditions.
2. Native aortic valve annulus size and morphology not suitable for Lotus or Sapien prosthesis implantation
3. Preexisting bioprosthetic valve or ring in aortic valve position.
4. Pre-existing pacemaker or ICD/CRT.
5. Cardiogenic shock or hemodynamic instability.
6. History of active endocarditis
7. Contraindications for a trans-femoral access.
8. Severe left ventricular dysfunction with LVEF <30%.
9. Severe mitral valve insufficiency.
10. Echocardiographic evidence of intracardiac mass, thrombus or vegetation.
11. Patients actively participating in another drug or device investigational study and have not yet completed the primary endpoint follow-up period.
12. Patients suffering from dementia.
13. Pregnant or nursing women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Incidence of new permanent pacemaker implantation | 30 days
  implantation of PM

SECONDARY OUTCOMES:
incidence of any prosthesis regurgitation | 30 days
  prosthesis regurgitation in echocardiography
Incidence of any conduction abnormalities | 30 days
  conduction abnormalities on rest ECG
Device success rate according to VARC-2 definition | 30 days
  combined endpoint
Mortality rate | 30 days
  all-cause death
Mortality rate | 1 year
  all-cause death
Mortality rate | 2 years
  all-cause death
incidence of early safety parameters according to VARC-2 definitions | 30 days
  combined endpoint
incidence of combined efficacy according to VARC-2 definitions | 1 year
  combined endpoint
incidence of combined efficacy according to VARC-2 definitions | 2 years
  combined endpoint

CONTACTS AND LOCATIONS:
Overall Officials: Julinda Mehilli, MD, Principal Investigator — Munich University Clinic, Ludwig-Maximilians University
Locations (3):
- Germany (2):
  - Munich University Clinic, Ludwig-Maximilians University, Munich, Bavaria
  - Segeberger Kliniken Gmbh, Bad Segeberg, Schleswig-Holstein
- Azienda Ospedaliero-Universitaria Pisana, Pisa, Italy

IPD SHARING:
Plan to Share IPD: No